CLINICAL TRIAL: NCT04627285
Title: A Multicenter, Open-Label, Follow-Up Study to Assess the Long-Term Use of Oral Lacosamide in Study Participants Who Completed EP0034 or SP848 and Received Lacosamide Treatment
Brief Title: A Study to Test the Long-term Use of Oral Lacosamide in Pediatric Study Participants Who Completed NCT01964560 (EP0034) or NCT00938912 (SP848) and Received Lacosamide Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EP0151; 2020-001478-30 (EudraCT Number); 2022-502639-21-00 (Registry Identifier: EU CT Number); U1111-1286-3095 (Other: Universal Trial Number (UTN))
Record Dates: First submitted 2020-11-12; First posted 2020-11-13 (Actual); Results first posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Epilepsy
Keywords: Lacosamide; Vimpat; Epilepsy; Pediatric
MeSH Terms: conditions — Epilepsy | interventions — Lacosamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Lacosamide (Experimental): Subjects in this arm will receive various single doses of lacosamide
  Interventions: Drug: Lacosamide

INTERVENTIONS:
Drug: Lacosamide — * Pharmaceutical form: Oral-solution
  * Route of administration: Oral use
  Subjects will receive lacosamide in a pre-specified sequence during the Treatment Period.

SUMMARY:
The purpose of the study is to assess the long-term use of lacosamide oral solution dosed at 2 mg/kg/day to 12 mg/kg/day when administered to pediatric study participants with epilepsy who have completed NCT01964560 (EP0034) or NCT00938912 (SP848).

ELIGIBILITY:
Inclusion Criteria:

* Participant is male or female, aged <6 years at the time of signing the Informed Consent Form (ICF)
* Participant has completed participation in NCT01964560 (EP0034) or NCT00938912 (SP848)
* Participant is expected to benefit from participation, in the opinion of the Investigator

Exclusion Criteria:

* Participant has any medical or psychiatric condition that, in the opinion of the Investigator, could jeopardize or would compromise the study participant's ability to participate in this study
* Participant has a known hypersensitivity to any components of the study medication or comparative drugs as stated in this protocol
* Participant is receiving any investigational drugs or using any experimental devices in addition to lacosamide (LCM)
* Participant meets a mandatory withdrawal criterion (ie, MUST withdraw criterion) for NCT01964560 (EP0034) or NCT00938912 (SP848), or is experiencing an ongoing serious adverse event (SAE)
* Sensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the Investigator or Medical Monitor, contraindicates participation in the study

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2020-12-28 (Actual); Primary Completion 2025-02-12 (Actual); Study Completion 2025-02-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (15):
- Georgia (3):
  - Ep0151 620, Tbilisi
  - Ep0151 621, Tbilisi
  - Ep0151 622, Tbilisi
- Hungary (2):
  - Ep0151 361, Budapest
  - Ep0151 362, Budapest
- Ep0151 650, Chisinau, Moldova
- Romania (3):
  - Ep0151 581, Bucharest
  - Ep0151 582, Iași
  - Ep0151 577, Timișoara
- Ep0151 224, Taipei, Taiwan
- Ukraine (5):
  - Ep0151 602, Dnipro
  - Ep0151 609, Dnipropetrovsk
  - Ep0151 606, Kiev
  - Ep0151 682, Uzhhorod
  - Ep0151 603, Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed.All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: https://www.Vivli.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll participants in December 2020 and concluded in February 2025.
Pre-assignment Details: Participants who completed studies EP0034 (NCT01964560) or SP848 (NCT00938912) were offered participation in this study. The Participant Flow refers to the Safety Set (SS).
Groups:
- Lacosamide: >=2 to <4 Years: Participants aged greater than or equal to (>=) 2 to less than (<) 4 years when entering EP0151 received LCM oral solution twice per day (BID) from a minimum dose of 2 milligram per kilogram per day (mg/kg/day) to a maximum dose of 12 mg/kg/day or 600 mg/day, to whichever was lower up to 209 weeks, based on optimization of seizure control and tolerability in the judgement of the Investigator.
- Lacosamide: >=4 to <6 Years: Participants aged >=4 to <6 years when entering EP0151 received LCM oral solution BID from a minimum dose of 2 mg/kg/day to a maximum dose of 12 mg/kg/day or 600 mg/day, to whichever was lower up to 209 weeks, based on optimization of seizure control and tolerability in the judgement of the Investigator.
Period: Overall Study
Arm/Group | Lacosamide: >=2 to <4 Years | Lacosamide: >=4 to <6 Years
Started | 19 | 29
Completed | 12 | 25
Not Completed | 7 | 4
Not completed — Adverse Event | 0 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Sponsor decision | 5 | 0
Not completed — Participant left country; aunt informed the site | 0 | 1

BASELINE CHARACTERISTICS:
Population: The SS consisted of all study participants who signed an informed consent form (ICF) and took at least 1 dose of study medication in this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lacosamide: >=2 to <4 Years | Lacosamide: >=4 to <6 Years | Total
Number analyzed (Participants) | 19 | 29 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 2.888 (0.518) | 5.180 (0.642) | 4.273 (1.277)
Age, Customized [Count of Participants; unit: Participants]
  Greater than or equal to (>=) 24 months to less than (<) 12 years | 19 | 29 | 48
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 15
  Male | 13 | 20 | 33
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 1 | 1 | 2
  Race: White | 18 | 28 | 46
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 0 | 3 | 3
  Ethnicity: Not Hispanic or Latino | 19 | 26 | 45

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An Adverse Event (AE) is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. Treatment-emergent AEs were defined as those events which started on or after the date of first dose of LCM in EP0151, or events for which severity worsened on or after the date of first dose of LCM in EP0151. Adverse events which occurred within 30 days after final dose of LCM in EP0151 were considered treatment-emergent.
Time Frame: From visit 1 (Week 0) to the end of study visit (up to Week 214.42)
Population: The SS consisted of all study participants who signed an ICF and took at least 1 dose of study medication in this study.
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide: >=2 to <4 Years | Lacosamide: >=4 to <6 Years
Number analyzed (Participants) | 19 | 29
percentage of participants | 42.1 | 37.9

2. Primary Outcome: Percentage of Participants Who Withdrew From Study Due to TEAEs
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. Treatment-emergent AEs were defined as those events which started on or after the date of first dose of LCM in EP0151, or events for which severity worsened on or after the date of first dose of LCM in EP0151. Adverse events which occurred within 30 days after final dose of LCM in EP0151 were considered treatment-emergent.
Time Frame: From visit 1 (Week 0) to the end of study visit (up to Week 214.42)
Population: The SS consisted of all study participants who signed an ICF and took at least 1 dose of study medication in this study.
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide: >=2 to <4 Years | Lacosamide: >=4 to <6 Years
Number analyzed (Participants) | 19 | 29
percentage of participants | 0.0 | 6.9

3. Primary Outcome: Percentage of Participants Who Withdrew From Study Due to Serious Adverse Event (SAEs)
Description: A SAE is defined as results in death, is life-threatening, requires in patient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly or birth defect, other important medical events which based on medical or scientific judgement may jeopardize the patients, or may require medical or surgical intervention to prevent any of the above. Only participants who discontinued the study due to SAEs are reported.
Time Frame: From visit 1 (Week 0) to the end of study visit (up to Week 214.42)
Population: The SS consisted of all study participants who signed an ICF and took at least 1 dose of study medication in this study.
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide: >=2 to <4 Years | Lacosamide: >=4 to <6 Years
Number analyzed (Participants) | 19 | 29
percentage of participants | 0.0 | 6.9

4. Primary Outcome: Modal Daily Dose During the Study
Description: The modal daily LCM dose in milligram per kilogram (mg/kg/day) is defined as the daily Lacosamide dose the participant received for the longest duration in EP0151.
Time Frame: From visit 1 (Week 0) to the end of study visit (up to Week 214.42)
Population: The SS consisted of all study participants who signed an ICF and took at least 1 dose of study medication in this study.
Measure: Mean (Standard Deviation); unit: mg/kg/day
Arm/Group | Lacosamide: >=2 to <4 Years | Lacosamide: >=4 to <6 Years
Number analyzed (Participants) | 19 | 29
mg/kg/day | 9.5 (2.4) | 10.0 (2.6)

5. Primary Outcome: Maximum Daily Dose During the Study
Description: Maximum daily dose is defined as the highest total daily dose a participant received in EP0151.
Time Frame: From visit 1 (Week 0) to the end of study visit (up to Week 214.42)
Population: The SS consisted of all study participants who signed an ICF and took at least 1 dose of study medication in this study.
Measure: Mean (Standard Deviation); unit: mg/kg/day
Arm/Group | Lacosamide: >=2 to <4 Years | Lacosamide: >=4 to <6 Years
Number analyzed (Participants) | 19 | 29
mg/kg/day | 9.5 (2.4) | 10.1 (2.6)

ADVERSE EVENTS:
Time Frame: From visit 1 (Week 0) to the end of study visit (up to Week 214.42)
Description: Treatment-emergent AEs were defined as those events which started on or after the date of first dose of LCM in EP0151, or events for which severity worsened on or after the date of first dose of LCM in EP0151. Adverse events which occurred within 30 days after final dose of LCM in EP0151 were considered treatment-emergent. Safety set included all participants who signed an ICF and took at least 1 dose of study medication.
Arm/Group | Lacosamide: >=2 to <4 Years | Lacosamide: >=4 to <6 Years
All-Cause Mortality (participants affected / at risk) | 0/19 | 2/29
Serious Adverse Events (participants affected / at risk) | 2/19 | 5/29
Other Adverse Events (participants affected / at risk) | 5/19 | 4/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lacosamide: >=2 to <4 Years (N=19) | Lacosamide: >=4 to <6 Years (N=29)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1)
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Device malfunction (General disorders) | 0 (0) | 1 (7)
Sudden death (General disorders) | 0 (0) | 1 (1)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia necrotising (Infections and infestations) | 0 (0) | 1 (1)
Rhinovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Partial seizures with secondary generalisation (Nervous system disorders) | 0 (0) | 1 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lacosamide: >=2 to <4 Years (N=19) | Lacosamide: >=4 to <6 Years (N=29)
Upper respiratory tract infection (Infections and infestations) | 5 (15) | 4 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-10-12): https://cdn.clinicaltrials.gov/large-docs/85/NCT04627285/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-08): https://cdn.clinicaltrials.gov/large-docs/85/NCT04627285/SAP_001.pdf